CLINICAL TRIAL: NCT04949139
Title: Efficacy and Safety of Rapid Intermittent Correction Compared With Slow Continuous Correction in Patients With Severe Hypernatremia (SALSA II Trial)
Brief Title: Efficacy and Safety of Rapid Intermittent Correction Compared With Slow Continuous Correction in Patients With Severe Hypernatremia
Acronym: SALSAII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-2104-680-003
Record Dates: First submitted 2021-06-06; First posted 2021-07-02 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-04

CONDITIONS: Hypernatremia
Keywords: Hypernatremia; Treatment; 5% dextrose water
MeSH Terms: conditions — Hypernatremia | interventions — Glucose; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rapid intermittent bolus group (Active Comparator): A : males < 65 ; B : females < 65 or males ≥ 65 ; C : females ≥ 65 yrs
  <During the first 3 h>
  Primary treatment over 1h A: 5DW 8 B: 5DW 7 C: 5DW 6 mL/kg
  If undercorrected, Repeat the 5DW amount infused during primary treatment after 3 h
  <At 3-24 h> Modify protocol based on sNa at each time point (6/12/18/24 h)
  Check U/S ratio at 0 h
  * undercorrection < 0.5: repeat the amount infused during primary treatment q 3 h
    ≥ 0.5: repeat the amount infused during primary treatment q 6 h
  * target correction < 0.5: repeat the amount infused during primary treatment q 6 h ≥ 0.5: stop the infusion
  <At 24-48 h> Modify protocol based on sNa at each time point (30/36/42/48 h)
  Check U/S ratio at 24 h
  * undercorrection < 0.5: repeat the amount infused during primary treatment q 3 h
    ≥ 0.5: repeat the amount infused during primary treatment q 6 h
  * target correction < 0.5: repeat the amount infused during primary treatment q 6 h ≥ 0.5: stop the infusion
  Interventions: Drug: Dextrose 5% in water
- Slow continuous infusion group (Active Comparator): Participants will be divided into three groups same as above
  <During the first 3 h>
  Primary treatment A: 5DW 1.8 B: 5DW 1.57 C: 5DW 1.35 mL/kg/h
  Modify protocol as described below based on sNa measurement at 3 h
  * undercorrection: maintain the infusion rate
  * target correction: stop the infusion
  <At 3-24 h> Modify protocol based on sNa measurement at each time point (6/12/18/24 h)
  Check U/S ratio at 0 h
  • undercorrection
  < 0.5: increase the infusion rate to twice that of the primary treatment
  ≥ 0.5: maintain the infusion rate
  • target correction
  < 0.5: maintain the infusion rate
  ≥ 0.5: stop the infusion
  <At 24-48 h> Modify protocol based on sNa measurement at each time point (30/36/42/48 h)
  Check U/S ratio at 24 h
  • undercorrection
  < 0.5: increase the infusion rate to twice that of the primary treatment
  ≥ 0.5: maintain the infusion rate
  • target correction
  < 0.5: maintain the infusion rate
  ≥ 0.5: stop the infusion
  Interventions: Drug: Dextrose 5% in water

INTERVENTIONS:
Drug: Dextrose 5% in water — Reducing the sodium concentration

SUMMARY:
This study will evaluate the efficacy and safety of rapid intermittent correction and slow correction with an electrolyte-free solution in patients with severe hypernatremia (glucose-corrected serum sodium, ≥ 155 mmol/L).

DETAILED DESCRIPTION:
Hypernatremia is defined as serum sodium (sNa) levels above 145 mmol/L and is caused by abnormalities in water balance, mainly in children, elderly, and critically ill patients. It occurs in 3% of hospitalized patients and in 9% of critically ill patients. Hypernatremia indicates hypertonic hyperosmolality and causes water outflow, resulting in cell dehydration. Most of the symptoms and signs of hypernatremia are due to brain abnormalities, which can progress to hyperventilation, muscle weakness, consciousness (lethargy), and coma. The short-term mortality rate of hypernatremia is 50%-60%. Decreased osmotic pressure in the extracellular fluid during correction of hyponatremia can cause cellular edema and permanent brain damage. The recommended sNa correction rate for acute hypernatremia is up to 1 mmol/L/h, whereas that for chronic hypernatremia is less than 0.5 mmol/L/h (approximately 10 mmol/L/day). However, these correction rates have only been studied and proven in pediatric patients. A recent study conducted on adults revealed that rapid correction (more than 0.5 mmol/L/h) was not associated with a higher risk for mortality, seizures, and alteration of consciousness. Several studies reported that excessively slow rates of sNa correction were associated with higher mortality, whereas rapid rates demonstrated lower mortality. There are no established guidelines for the Na correction rate for hypernatremia. The European and American guidelines recommend infusion of electrolyte-free water (10 mL/kg over 1 h or 3 mL/kg/h) for the management of overcorrection of hyponatremia. In the previously published SALSA I trial, 10 mL/kg over 1 h was applied as a method of re-lowering treatment in overly rapid correction of hyponatremia. However, this rapid intermittent bolus of electrolyte-free water has never been applied to treat hypernatremia.

The aim of this prospective, randomized, open-labeled, multi-center, and investigator-initiated trial is to determine whether a rapid and intermittent bolus of electrolyte-free water in hypernatremia can increase the incidence of rapid decrease in sNa level and increase the survival time compared to the slow continuous administration method. A total of 166 patients with severe hypernatremia will be enrolled and randomly assigned to receive either intermittent bolus or slow continuous infusion of 5% dextrose water. The participants will be divided into three groups according to age and sex and will receive 5% dextrose water for 2 days at different correction rates. Serum sodium will be measured every 3 h from the beginning to 6 h, followed by every 6 h until 48 h. In addition, urine sodium and potassium levels will be measured at baseline and 24 h. The PP (Per Protocol) analysis will be applied to enrolled participants who is infused with 75-125% of total planned volume of 5% dextrose water.

ELIGIBILITY:
Inclusion Criteria:

* Patients who visit the emergency department and in-patients over 18 years
* Severe hypernatremia: glucose-corrected serum sodium ≥ 155 mmol/L
* Written consent

Exclusion Criteria:

* Arterial hypotension requiring inotropes or vasopressors (systolic blood pressure < 90 mmHg and mean arterial pressure < 70 mmHg)
* Anuria or bilateral urinary outlet obstruction
* Uncontrolled diabetes mellitus (HbA1C > 9%) or glucose at baseline > 500 mg/dL or uncontrolled diabetic ketoacidosis or uncontrolled hyperosmolar hyperglycemic syndrome
* Decompensated liver cirrhosis (LC) - Known LC with ascites or diuretic use or hepatic encephalopathy or varix
* End-stage renal disease receiving renal replacement therapy
* Uncontrolled Heart failure (regardless of LVEF)
* Women who are pregnant or breast feeding
* Patients with the following conditions within 30 days prior to randomization:

  1. History of cardiac surgery excluding PCA, acute myocardial infarction, sustained ventricular tachycardia, ventricular fibrillation, acute coronary syndrome, and admission for heart failure
  2. Uncontrolled increase of intracranial pressure
* The subjects judged by investigators to have difficulty continuing the trial were also excluded.
* The case the subjects does not consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
efficacy : Incidence of rapid change in sNa level within 24 hours defined as follows | up to 24 hours
  Change in sNa by ≥ 6 mmol/L or Na ≤ 150 mmol/L within 24 hours All subjects will receive 5% dextrose water by rapid intermittent bolus or slow continuous infusion for 48 h, and sNa levels will be measured.

SECONDARY OUTCOMES:
the 28-day survival rate | up to 28 days
  survival rate
difference in sNa levels 6 hours after the initial test | up to 6 hours
  Gap of sodium level between 6 hours and initial level
volume of 5% dextrose water infused during 48 hours | up to 48 hours
  Volume
Incidence of rapid change in sNa level within 48 hours defined as follows | up to 48 hours
  Change in sNa by ≥ 12 mmol/L or Na ≤ 150 mmol/L within 48 hours

OTHER OUTCOMES:
Target correction rate | up to 48 hours
  Change in Na by ≥ 6 mmol/L and < 12 mmol/L from the initial level or Na ≤ 150 mmol/L within 24 hours Change in Na by ≥ 12 mmol/L and < 24 mmol/L from the initial level or Na ≤ 150 mmol/L within 48 hours
Incidence of undercorrection: | up to 48 hours
  sNa < 6 mmol/L within 3/6/12/24 hours sNa < 12 mmol/L within 48 h
Length of hospital stay | up to 8 weeks
  Length of hospital stay
Number of uses of desmopressin | up to 48 hours
  number of uses of demopressin
Incidence of overcorrection | up to 48 hours
  Na > 12 mmol/L within 24 h or > 24 mmol/L within 48 h at any given period
Incidence of cerebral edema documented via brain CT at 48 hours in patients with overcorrection | up to 48 hours
  incidence of cerebral edema
Incidence of osmotic demyelinating syndrome confirmed by ICD-10 code or MRI | up to 48 hours
  incidence of ODS
Glasgow coma scale at pretreatment, 6 hours, 24 hours, and 48 hours | up to 48 hours
  Glasgow coma scale can range from 3 (completely unresponsive) to 15 (responsive).
In-hospital mortality | up to 28 days
  mortality rate
Incidence of administrated intravenous volume of ≥ 3 L/day, except for fluids administrated according to the protocol | up to 48 hours
  incidence of adminitrated intravenous volume of ≥ 3 L/day

CONTACTS AND LOCATIONS:
Overall Officials: Sejoong Kim, PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qian Q. Hypernatremia. Clin J Am Soc Nephrol. 2019 Mar 7;14(3):432-434. doi: 10.2215/CJN.12141018. Epub 2019 Feb 6. No abstract available. PMID 30728169
- [Background] Chauhan K, Pattharanitima P, Patel N, Duffy A, Saha A, Chaudhary K, Debnath N, Van Vleck T, Chan L, Nadkarni GN, Coca SG. Rate of Correction of Hypernatremia and Health Outcomes in Critically Ill Patients. Clin J Am Soc Nephrol. 2019 May 7;14(5):656-663. doi: 10.2215/CJN.10640918. Epub 2019 Apr 4. PMID 30948456
- [Background] Hillier TA, Abbott RD, Barrett EJ. Hyponatremia: evaluating the correction factor for hyperglycemia. Am J Med. 1999 Apr;106(4):399-403. doi: 10.1016/s0002-9343(99)00055-8. PMID 10225241
- [Background] Adrogue HJ, Madias NE. Hypernatremia. N Engl J Med. 2000 May 18;342(20):1493-9. doi: 10.1056/NEJM200005183422006. No abstract available. PMID 10816188
- [Background] Sterns RH. Evidence for Managing Hypernatremia: Is It Just Hyponatremia in Reverse? Clin J Am Soc Nephrol. 2019 May 7;14(5):645-647. doi: 10.2215/CJN.02950319. Epub 2019 Apr 4. No abstract available. PMID 31064771
- [Background] Cabassi A, Tedeschi S. Severity of community acquired hypernatremia is an independent predictor of mortality: a matter of water balance and rate of correction. Intern Emerg Med. 2017 Oct;12(7):909-911. doi: 10.1007/s11739-017-1693-x. Epub 2017 Jul 1. No abstract available. PMID 28669048
- [Background] Lindner G, Funk GC. Hypernatremia in critically ill patients. J Crit Care. 2013 Apr;28(2):216.e11-20. doi: 10.1016/j.jcrc.2012.05.001. Epub 2012 Jul 2. PMID 22762930
- [Background] Bataille S, Baralla C, Torro D, Buffat C, Berland Y, Alazia M, Loundou A, Michelet P, Vacher-Coponat H. Undercorrection of hypernatremia is frequent and associated with mortality. BMC Nephrol. 2014 Feb 21;15:37. doi: 10.1186/1471-2369-15-37. PMID 24559470
- [Background] Alshayeb HM, Showkat A, Babar F, Mangold T, Wall BM. Severe hypernatremia correction rate and mortality in hospitalized patients. Am J Med Sci. 2011 May;341(5):356-60. doi: 10.1097/MAJ.0b013e31820a3a90. PMID 21358313
- [Background] Sterns RH, Silver SM. Salt and water: read the package insert. QJM. 2003 Aug;96(8):549-52. doi: 10.1093/qjmed/hcg102. No abstract available. PMID 12897339
- [Background] Spasovski G, Vanholder R, Allolio B, Annane D, Ball S, Bichet D, Decaux G, Fenske W, Hoorn EJ, Ichai C, Joannidis M, Soupart A, Zietse R, Haller M, van der Veer S, Van Biesen W, Nagler E; Hyponatraemia Guideline Development Group. Clinical practice guideline on diagnosis and treatment of hyponatraemia. Eur J Endocrinol. 2014 Feb 25;170(3):G1-47. doi: 10.1530/EJE-13-1020. Print 2014 Mar. PMID 24569125